CLINICAL TRIAL: NCT03079479
Title: Impact on Muscle Strength, Quality of Life and Functionality in Individuals Submitted to Hip Arthroplasty
Brief Title: Impact on Muscle Strength, Quality of Life and Functionality in Individuals Submitted to Hip Arthroplasty: a Prospective Study.
Status: Completed | Type: Observational
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, IMPACT ON MUSCLE STRENGTH, QUALITY OF LIFE AND FUNCTIONALITY IN INDIVIDUALS SUBMITTED TO HIP ARTHROPLASTY: A PROSPECTIVE STUDY, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: ccazarini
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2016-05

CONDITIONS: Arthroplasty Complications; Arthropathy of Hip
Keywords: Arthoplasty; Gait; muscle strenght; Quality of life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Two Years Group
  Interventions: Diagnostic Test: Muscle Strenght assesment; Diagnostic Test: 2D Kinematics Analysis
- Five Years Group
  Interventions: Diagnostic Test: Muscle Strenght assesment; Diagnostic Test: 2D Kinematics Analysis
- Ten Years Group
  Interventions: Diagnostic Test: Muscle Strenght assesment; Diagnostic Test: 2D Kinematics Analysis
- Control Group
  Interventions: Diagnostic Test: Muscle Strenght assesment; Diagnostic Test: 2D Kinematics Analysis

INTERVENTIONS:
Diagnostic Test: Muscle Strenght assesment — Muscle Strenght assesment of the hip muscles
Diagnostic Test: 2D Kinematics Analysis — 2D Kinematics Analysis of the gait

SUMMARY:
Introduction: Total hip arthroplasty has been increasingly used as a means of treating the various pathologies of this joint. However, this surgical reconstruction initially brings important deficits in subjects submitted, such as: inhibition of muscle strength, limitation of range of motion and functional deficit. Therefore, an immediate physiotherapeutic treatment is necessary in the short and long term, taking into account both biomechanical issues and the quality of life of these individuals.

Objective: To evaluate the clinical evolution of individuals submitted to total hip arthroplasty in the ten year period.

Method: Twenty individuals submitted to unilateral total hip arthroplasty will be evaluated by the medical group of hip surgeries of the Brotherhood of Santa Casa de Misericórdia of São Paulo, during a period of ten years. These individuals will undergo a primary clinical evaluation and after signing the consent form, will be evaluated functionally with the HARRIS HIP SCORE and WHOQOL-bref questionnaires and physically with the analysis of muscular strength through manual dynamometry to measure the strength level of the Muscles involved in the bilateral coxo-femoral joint, such as abductors, adductors, flexors, extensors, internal rotators, external rotators, knee joint, such as extensors and flexors, and ankle, plantar flexors. Finally, they will be referred to the kinematic gait analysis, to identify the functional characteristics of these individuals, through reflexive markers at specific anatomical points, where they will walk for 5 minutes on a treadmill at a speed of 1.5km per hour.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria in the study will be: patients submitted to total hip arthroplasty between 2 years (24 months - 35 months), 5 years (60 months - 71 months) and 10 years (120 months - 131 months), age between 50 and 80 years and sign the terms of free and informed consent

Exclusion Criteria:

* The exclusion criteria will be: patients with a history of prosthesis dislocations or revision of the arthroplasty, pain in the hip or lower limb region, asymmetry of the lower limbs greater than 2 centimeters, previous surgeries in the lower limbs, limitation of range of motion in the joint (Impossible to perform muscle strength tests), use of antidepressive drugs or analgesics of continuous use, chronic diseases not controlled (Hypertension, rheumatoid arthritis and diabetes) and the presence of neuromuscular pathologies

Ages: 56 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with total hip arthroplasty through the postero lateral approach
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Muscle strenght | Performed in a single evaluation
  Hand-Held dynamometer (Lafayette)

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Giannotti S, Bottai V, Dell'Osso G, De Paola G, Bugelli G, Guido G. The hip prosthesis in lateral femur fracture: current concepts and surgical technique. Clin Cases Miner Bone Metab. 2014 Sep;11(3):196-200. PMID 25568653
- [Result] Liu XW, Zi Y, Xiang LB, Wang Y. Total hip arthroplasty: areview of advances, advantages and limitations. Int J Clin Exp Med. 2015 Jan 15;8(1):27-36. eCollection 2015. PMID 25784971